CLINICAL TRIAL: NCT02439346
Title: An Open-label, Non-randomized, Multicenter Phase I Study to Characterize the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Maximum Tolerated Dose of Oral MKNK1 Inhibitor BAY 1143269 Given Alone or in Combination With Intravenous Docetaxel in Subjects With Advanced Solid Tumors
Brief Title: Phase I Dose Escalation and Expansion of Oral BAY 1143269 in Combination With Intravenous Docetaxel
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped due to project prioritization
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17450; 2014-004810-27 (EudraCT Number)
Record Dates: First submitted 2015-05-07; First posted 2015-05-08 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Medical Oncology
Keywords: Advanced solid tumors; Docetaxel; mitogen-activated protein (MAP) kinase-interacting serine / threonine-protein kinase 1, also known as Mnk1 (MKNK1 inhibitor); Taxanes; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BAY1143269 5 mg (Experimental): Subjects received BAY1143269 5 milligram (mg) tablet orally, once daily (QD) from Day 1 to 21 in treatment cycle until evidence of tumor progression, unacceptable toxicity, consent withdrawal, or withdrawal from the study at the discretion of the investigator. A treatment cycle consisted of 21 days.
  Interventions: Drug: BAY1143269 tablet
- BAY1143269 10 mg (Experimental): Subjects received BAY1143269 10 mg (2*5 mg) tablet orally, QD from Day 1 to 21 in treatment cycle until evidence of tumor progression, unacceptable toxicity, consent withdrawal, or withdrawal from the study at the discretion of the investigator. A treatment cycle consisted of 21 days.
  Interventions: Drug: BAY1143269 tablet
- BAY1143269 25 mg (Experimental): Subjects received BAY1143269 25 mg tablet orally, QD from Day 1 to 21 in treatment cycle until evidence of tumor progression, unacceptable toxicity, consent withdrawal, or withdrawal from the study at the discretion of the investigator. A treatment cycle consisted of 21 days.
  Interventions: Drug: BAY1143269 tablet
- BAY1143269 50 mg (Experimental): Subjects received BAY1143269 50 mg (2*25 mg) tablet orally, QD from Day 1 to 21 in treatment cycle until evidence of tumor progression, unacceptable toxicity, consent withdrawal, or withdrawal from the study at the discretion of the investigator. A treatment cycle consisted of 21 days.
  Interventions: Drug: BAY1143269 tablet

INTERVENTIONS:
Drug: BAY1143269 tablet — BAY 1143269 5 mg or 25 mg tablet. Each treatment cycle will last 21 days.

SUMMARY:
Determine the safety, tolerability, maximum tolerated dose (MTD), pharmacokinetics (PK), and/or recommended Phase II dose (RP2D) of oral BAY 1143269 given alone or in combination with intravenous (IV) docetaxel in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
BAY 1143269 is a potent and selective, orally administered novel inhibitor of mitogen-activated protein kinase interacting serine/threonine-protein kinase 1 (MKNK1). MKNK1 activity is essential for the phosphorylation of eukaryotic translation initiation factor 4E (eIF4E), which promotes the synthesis of oncogenic proteins, inhibits apoptosis, and helps tumor cells survive under stress. Increased p-EIF4E levels were found in tumor tissues from cancer patients. MKNK also functions as a mediator of pro-inflammatory cytokine production.

Established anti-mitotic drugs such as vinca alkaloids, taxanes, or epothilones activate the spindle assembly checkpoint (SAC), a key surveillance mechanism that monitors the attachment of spindle microtubules to the kinetochores of the chromosomes during pro-metaphase and halts the transitions to anaphase until all chromosomes are bi-oriented, fully attached, and correctly tensed at the metaphase plate. These antimitotic drugs destabilize or stabilize the spindle microtubules and cause mitotic arrest. Prolonged arrest in mitosis forces a cell either into a mitotic exit without cytokinesis or into a mitotic catastrophe leading to cell death. MKNK1 inhibitors allow cell apoptosis and increase tumor death. The combination of taxane and MKNK1 inhibitor can ultimately delay tumor progression and may provide a useful anticancer therapeutic approach.

This study will attempt to answer the following questions:

* What is the maximum tolerated dose (MTD) of BAY 1143269 when given alone or in combination with docetaxel?
* What is the safety profile and pharmacokinetics of BAY1143269 when given at the MTD?
* What are the adverse events of BAY 1161909 when given at different dose levels with docetaxel?

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged > 18 years
* Subjects must have histologically or cytologically confirmed locally advanced or metastatic solid tumors and must be refractory to any standard therapy, or have no standard therapy available, or have actively refused any standard therapy or, in the investigator's opinion, experimental treatment in this study is clinically and ethically acceptable for the subject.
* Subjects must have at least 1 measurable or evaluable tumor lesion according to RECIST 1.1 (Response Evaluation Criteria in Solid Tumors, version 1.1)
* Subjects must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Subjects must have a life expectancy of at least 12 weeks
* Subjects must have adequate bone marrow function as assessed by the following: hemoglobin >=9.0 g/dL or >=5.6 mmol/L, absolute neutrophil count (ANC) >=1.500/mm^3 or >=1.5 x 10^9/L (CTCAE Grade <=1), platelet count >= 100000/mm^3 or >=100 x 10^9/L
* Subjects must have adequate kidney function, as assessed by the estimated glomerular filtration rate (eGFR) >=60 mL/min per 1.73 m*2 [Common Terminology Criteria for Adverse Events(CTCAE Grade <=1)] calculated by the Modification of Diet in Renal Disease Study Group (MDRD) formula
* Subjects must have adequate liver function assessed by: total bilirubin <= 1.0 x upper limit of normal (ULN), aspartate aminotransferase (ALT) <= 3.0 x ULN (CTCAE Grade <=1) or, if receiving BAY1143269 in combination with IV docetaxel, AST and ALT <=1.5 x ULN if concomitant with alkaline phosphatase increase >2.5 x ULN
* Subjects must have adequate coagulation as assessed by: international normalized ratio (INR) or prothrombin time (PT) <=1.5 times ULN (CTCAE Grade <=1), partial thromboplastin time (PTT) <=1.5 x ULN (CTCAE Grade <=1)
* Women of reproductive potential must have a negative serum beta human chorionic gonadotropin (b-HCG) pregnancy test within 7 days before the first dose of study drug. Women of reproductive potential and men with female partners of childbearing potential must agree to consistently use highly effective contraception between signing the informed consent and 60 days after the last administration of study drug

Exclusion Criteria:

* Subjects who have a previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis) or any previous cancer curatively treated <3 years before the first dose of study drug
* Subjects who have a history of, or current evidence of bleeding disorder, i.e. any hemorrhage / bleeding event of CTCAE Grade >= 2 <4 weeks before the first dose of study drug.
* Subjects who have new or progressive brain or meningeal or spinal metastases
* Subjects who have a history of, or current evidence of uncontrolled cardiovascular disease or a left ventricular ejection fraction (LVEF) <50%
* Women who are pregnant or breast-feeding
* Subjects experiencing unresolved toxicity of previous antitumor therapy (excluding alopecia) which is CTCAE Grade >1 at screening
* Subjects who are current smokers or users of other tobacco products or have quit <90 days before first dose of study drug
* Subjects taking or likely to take strong and moderate CYP2D6 inhibitors, strong CYP1A1 inhibitors, and/or CYP1A1/CYP1A2 sensitive substrates or with narrow therapeutic index. Subjects receiving oral BAY1143269 and IV docetaxel must not take or be likely to take strong CYP3A1 inhibitors
* Subjects who have received systemic antitumor therapy within 4 weeks or radiotherapy to target lesions within 3 weeks before the first dose of study drug, which is longer
* Subjects who had received investigational drug treatment, including BAY1143269 and docetaxel, outside of this study within 4 weeks before the first dose of study drug, or for small molecules within the 5 half-lives of the agent before the first dose of study drug, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Oral BAY1143269 Alone and in Combination With Intravenous Docetaxel | Up to 2 years
  The MTD of oral BAY1143269 given alone was defined as the maximum dose at which the predicted incidence of dose-limiting toxicities (DLTs) during Cycle 1 is below 30 percent (%).
Maximum Observed Drug Concentration (Cmax) in Plasma After Single and Multiple Dose Administration of BAY1143269 | Cycle 1, 2 Day 1: Pre-dose to 24 hours post-dose
  Maximum observed concentration of BAY1143269 in plasma after single dose and multiple dose administration was measured.
Area Under the Concentration-time Curve From Time Zero to 24 Hours [AUC(0-24)] After Single and Multiple Dose Administration of BAY1143269 | Cycle 1, 2 Day 1: Pre-dose to 24 hours post-dose
  Area under the concentration-time curve from zero to 24 hours after single dose and multiple dose administration of BAY1143269 in plasma was measured.

SECONDARY OUTCOMES:
Tumor response | Baseline; end of Cycle 2
  Tumor response was assessed by Response Evaluation Criteria in Solid Tumors(RECIST V1.1). Evaluation of target lesions included CR(Disappearance of all target lesions),PR(at least a 30% decrease in sum of diameters of target lesions),PD:at least a 20% increase in sum of diameters of target lesions, taking smallest sum recorded as reference since treatment started or appearance of one or more new lesions) and Stable disease(SD:neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD).Evaluation of non-target lesions included CR(disappearance of all non-target lesions and normalization of tumor marker level),Non-CR/PD(Persistence of 1 or more non target lesions and/or maintenance of tumor marker level above normal limits) and PD(Appearance of 1 or more new lesions and/or unequivocal progression of existing non target lesions).

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (3):
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
- Sutton, Surrey, United Kingdom

REFERENCES:
- [Derived] Luo H, Huang S. Inhibition of MNK pathway sensitizes nasopharyngeal carcinoma to radiotherapy. Anticancer Drugs. 2024 Feb 1;35(2):155-162. doi: 10.1097/CAD.0000000000001542. Epub 2023 Sep 11. PMID 37694854